CLINICAL TRIAL: NCT07366502
Title: Comprehensive Hematological and Biochemical Comparison of Low-Dose Liposomal Iron Versus Standard-Dose Conventional Oral Iron in Iron Deficiency Anemia Following Sleeve Gastrectomy: A Prospective, Randomized Clinical Trial
Brief Title: Liposomal vs Conventional Oral Iron After Sleeve Gastrectomy
Acronym: anemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medeni Şermet (Other)
Responsible Party: Sponsor-Investigator, Medeni Şermet, assoc.prof., MD., Goztepe Prof Dr Suleyman Yalcın City Hospital
Organization: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-GOSEK-102
Record Dates: First submitted 2025-12-24; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: İron Deficiency Anemia; Liposomal Iron Replacement; Conventional Iron Replacement
Keywords: Iron deficiency anemia; Post-Bariatric surgery; Complications; Laparoscopic Sleeve Gastrectomy; Liposomal ıron; Conventional ıron
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Title: Liposomal Iron (Group LD) (Experimental): Participants with iron deficiency anemia after laparoscopic sleeve gastrectomy receiving oral liposomal iron.
  Interventions: Drug: Liposomal Iron
- Arm 2 Title: Conventional Iron (Group KD) (Active Comparator): Participants with iron deficiency anemia after laparoscopic sleeve gastrectomy receiving conventional oral ferrous iron preparations.
  Interventions: Drug: conventional oral iron

INTERVENTIONS:
Drug: Liposomal Iron — Oral liposomal iron capsules containing 17 iron per capsule, adminstered as 2 capsules daily, taken independently of meals for 6 months.
  Arms: Arm 1 Title: Liposomal Iron (Group LD)
Drug: conventional oral iron — oral ferrous iron preparations (ferrous sulfate, ferrous fumarate, or ferrous gluconate), each providing 100-200 mg elemental iron once daily, administered on an empty stomatch with 200 mg vitamin c for 6 months.
  Arms: Arm 2 Title: Conventional Iron (Group KD)

SUMMARY:
Low-dose liposomal iron (17-34 mg elemental/day) was compared with standard conventional oral iron (100-200mg elemental/day) in the treatment of iron deficiency anemia following sleeve gastrectomy. Liposomal iron provided superior hematological improvement and gastrointestinal tolerance.

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 65 years
* History of laparoscopic sleeve gastrectomy performed at least 6 months prior to enrollment
* Diagnosis of iron deficiency anemia, defined as:
* Hemoglobin <12 g/dL in women or <13 g/dL in men, and
* Serum ferritin <30 ng/mL or transferrin saturation (TSAT) <20%
* Mild to moderate anemia (hemoglobin ≥9 g/dL)
* Ability to take and swallow oral medications
* Willingness to participate and provide written informed consent Exclusion Criteria
* Active gastrointestinal disease (e.g., inflammatory bowel disease, peptic ulcer disease, or gastrointestinal bleeding)
* Chronic kidney disease with estimated GFR <30 mL/min/1.73 m²
* Use of oral or parenteral iron, vitamin B12, or folate supplementation within the previous 3 months
* Iron overload or hemochromatosis (serum ferritin >300 ng/mL)
* Known allergy or intolerance to iron preparations
* Active malignancy
* Pregnancy or breastfeeding
* Known hemoglobinopathies (e.g., thalassemia, sickle cell disease)
* Blood transfusion within the previous 1 month
* Cognitive or psychiatric disorder interfering with study participation or protocol adherence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin Level From Baseline to Week 24 | 24 weeks
  The change in hemoglobin concentration will be calculated as the absolute difference between baseline and week 24 values.

SECONDARY OUTCOMES:
Change in Serum Ferritin Level From Baseline to Week 24 | 24 weeks
  Absolute change in serum ferritin concentration from baseline to week 24.
Change in Transferrin Saturation (TSAT) From Baseline to Week 24 | 24 weeks
  Absolute change in transferrin saturation percentage from baseline to week 24.
Change in Serum Iron Level From Baseline to Week 24 | 24 weeks
  Absolute change in serum iron concentration from baseline to week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Prof.Dr. Suleyyman Yalçın City Hospital, Istanbul, kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We can share anonymized demographic and laboratory data upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38156148/

DOCUMENTS (1):
  • Study Protocol (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT07366502/Prot_000.pdf